CLINICAL TRIAL: NCT00924391
Title: Efficacy of Sterol Enhanced Soy Beverage on Cholesterol Metabolism, Inflammation and Oxidative Status in Humans Study 1
Brief Title: Efficacy of Sterol Enhanced Soy Beverage on Cholesterol Metabolism, Inflammation and Oxidative Status in Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: WhiteWave Foods, Inc. (Industry)
Responsible Party: Peter JH Jones, Richardson Centre for Functional Foods and Nutraceuticals
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: WWB2007:110
Record Dates: First submitted 2009-06-16; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Coronary Heart Disease
Keywords: cholesterol; plant sterols; cholesterol absorption
MeSH Terms: conditions — Coronary Disease | interventions — Milk

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- dairy milk (Active Comparator): Control phase with 1% milk.
  Interventions: Dietary Supplement: 1% milk
- phytosterol enhanced soy based beverage (Experimental): Treatment phase where control-phase diets are provided with phytosterol enhanced soy based beverage.
  Interventions: Dietary Supplement: phytosterol enhanced soy based beverage

INTERVENTIONS:
Dietary Supplement: phytosterol enhanced soy based beverage
  Arms: phytosterol enhanced soy based beverage
Dietary Supplement: 1% milk
  Arms: dairy milk

SUMMARY:
It is becoming increasingly clear that North Americans prefer dietary approaches to enhance health in favour of pharmaceutical approaches. Although the consumption of various phytosterol (PS)-enriched foods have been shown to be effective in lowering plasma cholesterol in a variety of food matrices, the lipid-lowering potential of PS-enriched soymilk has not been investigated. Therefore, the objective of this investigation was to examine the lipid-lowering efficacy of a PS-enriched soymilk beverage in comparison to a 1% dairy milk control. Twenty-three hypercholesterolemic subjects (Total-cholesterol and LDL-cholesterol ≥ 5.0 and 3.5 mmol/L, respectively) consumed 3 tetrapacs per day of a phytosterol-enriched soy beverage providing 1.95g PS/d or a 1% dairy milk control. The study was conducted as a 28 d controlled dietary intervention according to a completely randomized, two-period cross-over design.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, aged 19-60 yr, will be screened for determination of fasting circulating LDL-cholesterol and TG levels.
2. Subjects accepted into the study will have plasma LDL-C 130-200 mg/dl, TG levels below 250 mg/dl.
3. The inclusion for body mass index (BMI) range will be 22 to 32 kg/m2.
4. Subjects must also demonstrate an ability to understand dietary procedures and exercise procedures and be judged as compliant and motivated by the investigators.
5. Subjects will be permitted to take stable doses of thyroid hormone and anti-hypertensive agents, as long as these are continued equivalently throughout the duration of study.

Exclusion Criteria:

1. History of recent (i.e. less than 3 months) or chronic use of oral hypolipidemic therapy, including fish oils, or probucol within the last 6 months.
2. History of chronic use of alcohol (> 2 drinks/day), systemic antibodies, corticosteroids, androgens, or phenytoin.
3. Myocardial infarction, coronary artery bypass, or other major surgical procedures within the last six months.
4. Recent onset of angina, congestive heart failure, inflammatory bowel disease, pancreatitis, diabetes, or significant current (ie. onset within past three months) gastrointestinal, renal, pulmonary, hepatic or biliary disease, or cancer (evidence of active lesions, chemotherapy or surgery in the past year).
5. Exercise greater than 15 miles/wk or 4,000 kcal/wk.

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2007-09; Primary Completion 2007-12 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
cholesterol | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter JH Jones, B.ScM.ScPh.D, Principal Investigator — Richardson Centre for Functional Foods and Nutraceuticals
Locations (1):
- Richardson Centre for Functional Foods and Nutraceuticals, Winnipeg, Manitoba, Canada

REFERENCES:
- [Derived] Rideout TC, Chan YM, Harding SV, Jones PJ. Low and moderate-fat plant sterol fortified soymilk in modulation of plasma lipids and cholesterol kinetics in subjects with normal to high cholesterol concentrations: report on two randomized crossover studies. Lipids Health Dis. 2009 Oct 20;8:45. doi: 10.1186/1476-511X-8-45. PMID 19843338